CLINICAL TRIAL: NCT03680547
Title: Pattern of Sickle Cell Nephropathy in Patients With Sickle Cell Disease
Brief Title: Nephropathy in Patients With Sickle Cell Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, omnia talat hasan, assiut, Assiut University
Other Study IDs: npscd
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Sickle Cell Nephropathy
MeSH Terms: interventions — Hemoglobin, Sickle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient with sickle cell disease — assess degree of renal affection in patientswith sickle cell disease attending Assuit university Children hospital by estimating some predictors of glomerular and tubular dysfunction.

SUMMARY:
There are some diseases that give rise to diverse renal manifestations as does sickle cell disease

DETAILED DESCRIPTION:
Such involvement adversely affects virtually all major physiological processes in the kidney, and leads to complications that are common and chronic on the one hand (such as impaired urinary concentrating ability), and those that are rare and uniformly fatal on the other (such as renal medullary carcinoma) This steady adverse renal sequelae shortens the average lifespan of patients with SCD.

Proteinuria and a reduced glomerular filtration rate are risk factors associated with increased mortality among those patients with approximately 16-18% of overall mortality in this patient group is due to kidney disease.

Once end stage renal disease is reached, the mortality of patients who are on haemodialysis and have SCD is increased severalfold relative to the mortality of patients who are on haemodialysis but do not have SCD.

Thus,although the average lifespan of patients with SCD has increased during recent decades owing to improved management of complications outside the kidney,kidney disease contributes substantially to the still increased mortality in SCD.

ELIGIBILITY:
Inclusion Criteria:

* All patients with sickle cell anemia attending the unit will be included in the study.

Exclusion Criteria:

* patient with any underlaying systemic diseases other than sickle cell anaemia

Ages: 5 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: to assess degree of renal affection in patients with sickle cell disease attending Assuit university Children hospital by estimating some predictors of glomerular and tubular dysfunction.detailed history taking and thorough clinical examination and laboratory investigations
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
sickle cell nephropathy in patient with sickle cell disease | one year
  detection of renal impairment in patients with sickle cell disease by estamating gloerular and tubular dysfunction clinicaly and laboratory

CONTACTS AND LOCATIONS:
Overall Officials: omnia talat hasan, Principal Investigator — assiut

IPD SHARING:
Plan to Share IPD: Undecided